CLINICAL TRIAL: NCT00891813
Title: Effectiveness and Safety of a 6-Month Treatment With IV Zemplar in Patients on Hemodialysis and With Secondary Hyperparathyroidism Using iPTH/100 as Initial Dose
Brief Title: Effectiveness and Safety of IV Zemplar in Patients on Hemodialysis and With Secondary Hyperparathyroidism Using iPTH/100 as Initial Dose
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: W10-677
Record Dates: First submitted 2009-04-29; First posted 2009-05-01 (Estimated); Results first posted 2011-10-31 (Estimated); Last update posted 2011-10-31 (Estimated); Status verified 2011-09

CONDITIONS: Secondary Hyperparathyroidism; Renal Insufficiency, Chronic; Parathyroid Hormone; Hemodialysis; Hypercalcemia
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Renal Insufficiency, Chronic; Hypercalcemia | interventions — paricalcitol

ARMS (1):
- Zemplar (paracalcitol) (Experimental)
  Interventions: Drug: Zemplar (paricalcitol)

INTERVENTIONS:
Drug: Zemplar (paricalcitol) — Zemplar (paricalcitol) dose will be calculated mcg=PARATHYROID HORMONE level/100; this will be provided 3 times per week. Dose will be adjusted by 2-4 mcg every 4 weeks according to the parathyroid hormone level.
  Other Names: ABT-358; paricalcitol; Zemplar

SUMMARY:
The purpose of this study is to observe the effectiveness and safety of the use of a low initial dose regime (iPTH/100) in chronic kidney disease patients with secondary hyperparathyroidism (PTH>300pg/mL) and that require dialysis at least 3 times per week.

DETAILED DESCRIPTION:
The study will be carried out in three dialysis centers in Peru. Each patient enrolled in the study will be followed during a 6 month period from the time of inclusion. Study visits will occur at Baseline and at Weeks 4, 8, 12 and 24 during the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients >=18 years old with secondary hyperparathyroidism (PTH>300pg/mL, measured in the last 2 weeks).
* Patients on hemodialysis who require starting therapy with IV paricalcitol (de novo).
* Patients attending 3 hemodialysis sessions per week.
* Patients signing the informed consent approved by the Ethics Committee. If any individual is not capable of giving his/her consent, it can be obtained from a next of kin or from his/her legal representative, according to local laws and regulations.
* The decision to initiate treatment is upon the investigator and the decision to treat patients with IV paricalcitol must not be based on the inclusion of the patient in the study or any other way. The decision to treat a patient with IV paricalcitol will be taken prior to asking the patient to participate in the study.

Exclusion Criteria:

* Patients with any concomitant clinical condition that, according to the investigator's opinion, might impede an adequate assessment of the treatment response.
* Patients with severe hyperparathyroidism (PTH>3000pg/mL).
* Patients with a serum calcium level greater or equal to 10.5mg/dL, phosphorus greater or equal to 6.5mg/dL, or those with Calcium X Phosphorus product 65 (measured at least 2 weeks before the study).
* Patients with neoplastic disease.
* Pregnant or lactating women.
* Known hypersensitivity and/or toxicity to vitamin D metabolites and/or to other ingredients of the product.
* Having participated in another study with an investigational product or device within the previous 30 days or having planned to participate in another study within the same period of time as the actual study.
* Use of vitamin D analogue during the last 3 months prior to the inclusion to this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-05; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oscar E Guerra, MD, Study Director — Abbott
Locations (3):
- Peru (3):
  - Site Reference ID/Investigator# 21401, Callao
  - Site Reference ID/Investigator# 23857, Lima
  - Site Reference ID/Investigator# 10941, Lima

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 114 participants were screened. Of those, 100 participants were enrolled and received at least one dose of study drug.
Groups:
- Paricalcitol Injection: Initial dosage was calculated based on intact parathyroid hormone (iPTH) as follows: iPTH level/100 = micrograms (mcg) dose. Drug was administered 3 times per week. Dosage could be adjusted by 2 to 4 mcg every 4 weeks based on the participant's iPTH, calcium and phosphorus levels.
Period: Overall Study
Arm/Group | Paricalcitol Injection
Started | 100
Completed | 88
Not Completed | 12
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 1
Not completed — Patient Noncompliance | 6
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Arm/Group | Paricalcitol Injection
Number analyzed (Participants) | 100
Age Continuous [Mean (Standard Deviation); unit: years] | 46 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 53
Region of Enrollment [Number; unit: participants]
  Peru | 100

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Patients Reaching at Least a 30% Reduction in PTH and/or Values in Range 150-300 pg/mL
Description: The percentage of participants who achieved at least a 30% reduction in intact parathyroid hormone (iPTH) and/or an iPTH value in the range of 150 to 300 picograms per milliliter (pg/mL) at any post-baseline visit during the study. An iPTH value of 150-300 pg/ml is the target range recommended by the NKF KDOQI (National Kidney Foundation Kidney Disease Outcomes Quality Initiative) for End Stage Renal Disease patients.
Time Frame: 24 weeks
Population: Analysis is based on the number of participants completing the study.
Measure: Number; unit: Percentage of participants
Arm/Group | Paricalcitol Injection
Number analyzed (Participants) | 88
Percentage of participants | 96.6

2. Secondary Outcome: Time to Reach the First 30% Reduction in PTH and/or a Value Between 150-300pg/mL
Description: Median time to achieve at least a 30% reduction in intact parathyroid hormone (iPTH) and/or an iPTH value in the range of 150-300 pg/mL.
Time Frame: 24 Weeks
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | Paricalcitol Injection
Number analyzed (Participants) | 100
Weeks | 4 [2 to 6]

3. Secondary Outcome: Number of Participants With Hypercalcemia (>10.5mg/dL), Hyperphosphatemia (>6.5mg/dL) and/or Elevations of the Ca X P Product (>65).
Description: The number of participants with hypercalcemia (defined as at least one calcium value of more than 10.5 milligrams per deciliter [mg/dL]), hyperphosphatemia (phosphorus value of more than 6.5 mg/dL), and/or elevation of Calcium X Phosphorus product (value greater than 65) during the 24 week study.
Time Frame: 24 Weeks
Measure: Number; unit: Number of participants
Arm/Group | Paricalcitol Injection
Number analyzed (Participants) | 100
Number of participants
  Hypercalcemia | 38
  Hyperphosphatemia | 33
  Elevation of Ca x P product | 31

ADVERSE EVENTS:
Time Frame: Baseline through 24 weeks.
Description: The investigators monitored each participant for clinical and laboratory evidence of adverse events on a routine basis throughout the study. All serious and non serious adverse events from the time participant received the first dose of study drug until one month after the last dose of paricalcitol were reported.
Arm/Group | Paricalcitol Injection
Serious Adverse Events (participants affected / at risk) | 15/100
Other Adverse Events (participants affected / at risk) | 47/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paricalcitol Injection (N=100)
Acute coronary syndrome (Cardiac disorders) | 1
Atrioventricular block complete (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 2
Cellulitis (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 5
Humerus fracture (Injury, poisoning and procedural complications) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Paricalcitol Injection (N=100)
Hypercalcemia (Metabolism and nutrition disorders) | 32
Hyperphosphatemia (Metabolism and nutrition disorders) | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.